CLINICAL TRIAL: NCT03962907
Title: Preoperative Decolonization and Surgical Site Infections in Orthopaedic Surgery: a Prospective Randomized Controlled Trial - 2 Year Outcome in Prosthetic Surgery
Brief Title: Preoperative Decolonization and Surgical Site Infections in Orthopaedic Surgery - 2 Year Outcome in Prosthetic Surgery
Acronym: DECO-SSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lindenhofgruppe AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DECO-SSI P 2
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2019-10

CONDITIONS: Staphylococcus Aureus; Orthopaedic Surgery; Surgical Site Infection; Prevention
MeSH Terms: conditions — Staphylococcal Infections; Surgical Wound Infection | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: two groups: S. aureus carrier and non-carriers. Both groups have an intervention and control arm
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are not told colonization status or study arm. Outcome Assessor are not informed as well on this informations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Carrier group - intervention (Experimental): BACTROBAN® Nasal ong, 3g, GSK Lifo-Scrub sol 4%®, 500ml, B. Braun
  Interventions: Drug: Chlorhexidine, Lifo-Scrub sol 4%®, 500ml, B. Braun; Drug: BACTROBAN® Nasal ong
- Carrier group - control (No Intervention)
- Non - carrier group - intervention (Experimental): Lifo-Scrub sol 4%®, 500ml, B. Braun
  Interventions: Drug: Chlorhexidine, Lifo-Scrub sol 4%®, 500ml, B. Braun
- Non - carrier group - control (No Intervention)

INTERVENTIONS:
Drug: Chlorhexidine, Lifo-Scrub sol 4%®, 500ml, B. Braun — 5 - day decolonization procedure prior elective surgery. In carriers with Chlorhexidine daily showers and Mupirocin twice a day nasal ointment. In non-carriers Chlorhexidine showers will be used.
  Arms: Carrier group - intervention; Non - carrier group - intervention
Drug: BACTROBAN® Nasal ong — Mupirocin, BACTROBAN® Nasal ong, 3g, GSK
  Arms: Carrier group - intervention

SUMMARY:
Surgical site infections in orthopaedic surgery are a major problem. Decolonization has been suggested to reduce infection rates. The study was designed as a prospective, controlled, randomized, single-blinded trial to assess the influence of a decolonization procedure in S. aureus and non - S. aureus carriers. In this trial the 2 - year outcome in the subpopulation of prosthetic elective orthopaedic surgery will be evaluated.

DETAILED DESCRIPTION:
To verify the main hypothesis, a prospective controlled randomized interventional trial with 2 parallel groups of patients of the Sonnenhof hospital undergoing an elective knee- or hip implant surgery was designed. A superiority framework for the decolonization procedure was used. All patients planned for such a procedure will be recruited during preoperative consultation by the orthopedic surgeons or by post and phone. Written informed consent will be obtained at this occasion. Study participants were screened 2-4 weeks prior intervention for nasal S. aureus colonization.

Study participants were allocated on a 1:1 basis either to an intervention or to a control group, but prosthesis implantation was not defined as randomization criteria in the initial trial. Randomization was stratified for important risk factors of SSI; procedure type (upper extremities and pelvic/hip, spine, knee and foot) and ASA-criteria (I, II, III -V). Stratification-groups were chosen in function of SSI's rate and expected number of operations/year. Randomization list were generated by the CTU and allocation was concealed using central randomization that was implemented in the REDCap data entry system.

One week prior to hospitalization patients in the intervention group received a decolonization kit by mail with instructions to apply mupirocin ointment 2% (BACTROBAN Nasal ong 3g, GSK) in each nostril 30mg (which corresponds approximately the same amount as the volume of a pea) twice a day and to shower daily (starting with the face, then from top to bottom the whole body emphasizing especially on nose, axillaries and pelvic region and then rinse. In a second time starting with the hair and then repeat the whole body. Dry with a proper towel (one for the 5 days)) with 25ml chlorhexidine gluconate soap, (Lifo-Scrub sol 4 % 500ml, B. Braun) during 5 days prior surgery. For non S. aureus carriers only skin cleansing without intranasal mupirocin application was used. This dosing schedule, mode of administration and treatment periods correspond to the allowed and recommended standards of Swissmedic and were not modified in this trial. Decolonization occured before hospitalization, as a fully completed course before surgery has been more effective. In some of the previous trials decolonization took place only at the beginning of hospitalization. The decolonization procedure was only completed after surgery had taken place and this possibly affected the results.

For practical reasons the use of a placebo kit within the control group abandoned. Operators, who are also the outcome assessors, will be blinded for either the carrier status or the decolonization procedure. Study participants will be told not to inform surgeons about performed decolonization procedure.

The incidence of PJI at two years in the intervention and control group will be assessed by phone interview.

ELIGIBILITY:
Inclusion Criteria:

* older than 16 years
* planned elective orthopedic procedure
* Decolonization protocol can be performed timely

Exclusion Criteria:

* No orthopedic prosthetic surgery planned
* Allergy to mupirocin or chlorhexidine
* Presence of a nasal foreign body
* No informed consent
* undergoing treatment/surgery for a documented infection
* already participating in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1318 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Surgical site infections | 2 years
  according CDC-Criteria

SECONDARY OUTCOMES:
Overall mortality | 2 years
Death related to infection | 2 years
Documented bacteria | 2 years
  of PJI
Time to PJI and death | 2 years
  counting from operation date

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brügger, MD, Principal Investigator — Lindenhofgruppe
Locations (1):
- Sonnenhofspital, Lindenhofgruppe, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No